CLINICAL TRIAL: NCT00101673
Title: Efficacy and Safety of Vildagliptin in Patients With Type 2 Diabetes With HbA1c 9-11%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2329
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
This study was not conducted in the United States. The purpose of this study was to assess the safety and effectiveness of two doses of vildagliptin, an unapproved drug, in lowering overall blood glucose levels in people with type 2 diabetes who had not previously been treated with drug therapy to lower their blood sugar and whose blood sugar levels were in a specified range.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose criteria must be met
* Not currently on drug therapy for type 2 diabetes
* Body mass index (BMI) in the range 22-45

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* Evidence of serious diabetic complications
* Evidence of serious cardiovascular conditions
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2004-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 12 weeks

SECONDARY OUTCOMES:
Adverse event profile after 12 weeks of treatment
Patients with reduction in HbA1c >/= 0.7% after 12 weeks
Change from baseline in fasting plasma glucose at 12 weeks
Change from baseline in HOMA-B at 12 weeks
Change from baseline in body weight at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Pratley RE, Schweizer A, Rosenstock J, Foley JE, Banerji MA, Pi-Sunyer FX, Mills D, Dejager S. Robust improvements in fasting and prandial measures of beta-cell function with vildagliptin in drug-naive patients: analysis of pooled vildagliptin monotherapy database. Diabetes Obes Metab. 2008 Sep;10(10):931-8. doi: 10.1111/j.1463-1326.2007.00835.x. Epub 2007 Dec 17. PMID 18093207
- [Derived] Pratley RE, Rosenstock J, Pi-Sunyer FX, Banerji MA, Schweizer A, Couturier A, Dejager S. Management of type 2 diabetes in treatment-naive elderly patients: benefits and risks of vildagliptin monotherapy. Diabetes Care. 2007 Dec;30(12):3017-22. doi: 10.2337/dc07-1188. Epub 2007 Sep 18. PMID 17878242